CLINICAL TRIAL: NCT04387994
Title: Early Prediction of First Trimester Miscarriage After IVF With Serum Circulating Placental Biomarkers: a Pilot Study to Develop a Prediction Model.
Brief Title: Determination of Circulating Placental Biomarkers Levels to Predict the Pregnancy Outcome of First Trimester After IVF.
Status: Completed | Type: Observational
Sponsor: Instituto Valenciano de Infertilidade de Lisboa (Network)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor
Other Study IDs: 1812-LIS-104-TS
Record Dates: First submitted 2020-05-11; First posted 2020-05-14 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Infertility, Female; First Trimester Spontaneous Abortion
Keywords: Placental biomarkers; In vitro fertilization (IVF); Pregnancy outcome; Miscarriage; Early prediction; Intracytoplasmatic sperm injection (ICSI)
MeSH Terms: conditions — Infertility, Female; Abortion, Spontaneous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will be collected to determine the circulating placental biomarkers concentrations.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Blood samples collection — Collection of blood samples from consenting subjects to evaluate circulating biomarkers concentrations.

SUMMARY:
This study will assess the predictive potential of circulating placental biomarkers for spontaneous miscarriage within the following month in an IVF setting. It is hypothesized that a robust algorithm including one or more of these biomarkers may allow for the accurate same-day distinction between women with a low and high risk of a spontaneous miscarriage.

DETAILED DESCRIPTION:
Spontaneous miscarriage is the most common adverse outcome in the first trimester of pregnancy. This is a particularly stressful situation for the expecting parents, since their need for a final diagnosis is frustrated for a potentially extended period on time which may span over several weeks. The emotional impact of this complication can be devastating, resulting frequently in depression and anxiety which may last for several months.

In an attempt to allow for an earlier and more accurate diagnosis of first trimester miscarriage, multiple circulating placental biomarkers have been tested over last years. However, their potential usefulness in an everyday clinical setting remains unclear.

The investigators propose a single-center observational prospective cohort study in an in vitro fertilization (IVF) setting. All recruited consenting patients will collect blood samples on a day of the first pregnancy test (12-14 days after embryo transfer) and at the time of the first (at 5 weeks plus 4-5 days of gestational age) and second (at 7 weeks plus 4-5 days of gestational age) ultrasound scan to determine the circulating placental biomarkers concentrations in order to predict the pregnancy outcome (spontaneous miscarriage versus evolutive pregnancy) until the first obstetrical ultrasound, performed between 11 weeks and 13 weeks plus 6 days of gestational age.

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥18 and <49 years old
* Body Mass Index (BMI): ≥18.5 Kg/m2 and <30 Kg/m2
* Pregnancy resulting from Assisted Reproductive Technologies (ART)
* Single blastocyst transfer pregnancy
* Pregnancy confirmed by blood test
* Gestational age < 6 weeks at the first US
* Signed and dated informed consent

Exclusion Criteria:

* Spontaneous pregnancies
* Treatment for prevention of miscarriage (i.e. corticoids, aspirin, heparin)
* Those unable to provide the 11th-13th week ultrasound report
* Those unable to comprehend the investigational nature of the proposed study

Ages: 18 Years to 48 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: 120 pregnant subjects, confirmed by blood βhCG test, following vitrified-warmed single blastocyst cycles performing IVF/Intracytoplasmic Sperm Injection (ICSI) with autologous oocytes without preimplantation genetic testing for aneuploidies (PGT-A).
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2020-06-12 (Actual); Primary Completion 2021-12-07 (Actual); Study Completion 2021-12-07 (Actual)

PRIMARY OUTCOMES:
Pregnancy outcome (spontaneous miscarriage versus evolutive pregnancy) at the first trimester ultrasound | Up to the first trimester ultrasound (11 to 13 weeks plus 6 days of gestation)
  Measurement of circulating placental biomarkers levels

SECONDARY OUTCOMES:
Abnormal outcomes of early pregnancy (biochemical pregnancy and extra uterine pregnancy) | Up to the first trimester ultrasound (11 to 13 weeks plus 6 days of gestation)
  Measurement of circulating placental biomarkers levels
Risk of obstetric complications/adverse outcomes for first-trimester spontaneous miscarriage | Up to the first trimester ultrasound (11 to 13 weeks plus 6 days of gestation)
  Measurement of circulating placental biomarkers levels

CONTACTS AND LOCATIONS:
Overall Officials: Tetyana Semenova, MD, Principal Investigator — Instituto Valenciano de Infertilidade de Lisboa
Locations (1):
- Instituto Valenciano de Infertilidade de Lisboa, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: No